CLINICAL TRIAL: NCT01755143
Title: CapSureFix® Novus Model 5076 Lead MRI Study
Brief Title: Evaluation of Approved Pacing Lead (Model 5076) for Use in MRI Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 5076 MRI
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-06

CONDITIONS: Magnetic Resonance Imaging (MRI); Cardiac Pacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MRI Group (Experimental): Subjects randomized to the Magnetic Resonance Imaging group will undergo a series of MRI scans at the 9-12 week visit post-implant.
  Interventions: Other: Magnetic Resonance Imaging scan sequences of the head, neck, and chest; Device: Pacemaker System
- Control Group (Sham Comparator): Subjects randomized to the control group will not undergo a series of MRI scans but will come into the study office for a one hour waiting period at the 9-12 week post-implant visit.
  Interventions: Device: Pacemaker System

INTERVENTIONS:
Other: Magnetic Resonance Imaging scan sequences of the head, neck, and chest
  Arms: MRI Group
Device: Pacemaker System
  Other Names: Model 5076 Lead; Advisa MRI Pacemaker

SUMMARY:
The purpose of this study is to test the safety and effectiveness of the Medtronic CapSureFix Novus Model 5076 lead when patients are implanted with the Medtronic Advisa MRI pacemaker and undergo an MRI scan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have Class I and II indication for implantation of a dual chamber pacemaker according to the ACC/AHA/HRS guidelines
* Subjects who are able to undergo a pectoral implant
* Subjects who:
* are receiving an IPG for the first time, OR
* are receiving a replacement IPG connected to two previously- implanted (atrial and ventricular) Model 5076 leads
* Subjects who are able and willing to undergo elective MRI scanning without sedation
* Subjects who are geographically stable and available for follow-up at the study site for the length of the study

Exclusion Criteria:

* Subjects with a mechanical tricuspid heart valve.
* Subjects with a history of significant tricuspid valvular disease.
* Subjects for whom a single dose of 1.0mg dexamethasone acetate may be contraindicated.
* Subjects who require a legally authorized representative to obtain consent.
* Subjects who have abandoned (inactive) pacemaker and/or defibrillator leads
* Subjects who are immediate candidates for an ICD.
* Subjects who require an indicated MRI scan, other than those specifically described in the study, before the one-month post MRI/waiting period follow-up.
* Subjects with previously implanted active medical devices (exception Model 5076 Lead and Advisa MRI IPG).
* Subjects with a non-MRI compatible device (such as ICDs or neurostimulators) or material implant (e.g., non-MRI compatible sternal wires, neurostimulators, biostimulators, metals or alloys).
* Subjects with medical conditions that preclude the testing required by the protocol or limit study participation.
* Subjects who are enrolled or intend to participate in another clinical trial (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during this clinical study.
* Pregnant women, or women of child bearing potential and who are not on a reliable form of birth control.
* Subjects with exclusion criteria required by local law (e.g., age, breastfeeding).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2012-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- Australia (2):
  - Saint George Hospital, Kogarah, New South Wales
  - Flinders Medical Centre, Bedford Park
- Austria (2):
  - Landesklinikum St. Pölten, Sankt Pölten
  - Wilhelminenspital, Vienna
- Belgium (2):
  - Les Cliniques du Sud Luxembourg Cliniques Saint Joseph, Arlon
  - Hôpital Saint-Joseph, Gilly
- Hospital Clínico Pontificia Universidad Católica, Santiago, Chile
- Prince of Wales Hospital Hong Kong, Hong Kong, China
- Fundacion Cardioinfantil, Bogotá, Colombia
- Germany (4):
  - Klinikum Links der Weser, Bremen
  - Praxisklinik Herz und Gefässe, Dresden
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Ulm, Ulm
- Queen Mary Hospital, Hong Kong, Hong Kong
- India (7):
  - Medanta The Medicity, Gurgaon, Haryana
  - Sri Jayadeva Institute of Cardiovascular Sciences and Research, Bangalore
  - Post Graduate Institute of Medical Education & Research, Chandigarh
  - Fortis Escorts Hospital, Jaipur
  - Holy Family Hospital, Mumbai
  - All India Institute of Medical Sciences, New Delhi
  - Dayanand Medical College, Punjab
- Netherlands (3):
  - St. Antonius Ziekenhuis - Locatie Nieuwegein, Nieuwegein
  - Maasstad Ziekenhuis, Rotterdam
  - HagaZiekenhuis - Locatie Leyweg, The Hague
- Centro Hospitalar do Porto, Porto, Portugal
- Prince Sultan Cardiac Center, Riyadh, Saudi Arabia
- Serbia (2):
  - Klinicki Centar Srbije, Belgrade
  - Institut za Kardiovaskularne Bolesti Vojvodine, Kamenitz
- National Heart Centre Singapore, Singapore, Singapore
- Narodny ustav srdcovych a cievnych chorob, Bratislava, Slovakia
- Netcare Unitas Hospital, Pretoria, South Africa
- Hospital Universitari Clínic de Barcelona, Barcelona, Spain
- Switzerland (2):
  - HFR Fribourg - Hôpital cantonal, Fribourg
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- MRI Group: Subjects randomized to the Magnetic Resonance Imaging group will undergo a series of MRI scans at the 9-12 week visit post-implant.
  Magnetic Resonance Imaging scan sequences of the head, neck, and chest
  Pacemaker System
- Control Group: Subjects randomized to the control group will not undergo a series of MRI scans but will come into the study office for a one hour waiting period at the 9-12 week post-implant visit.
  Pacemaker System
Period: Overall Study
Arm/Group | MRI Group | Control Group
Started | 177 | 89
Completed | 166 | 86
Not Completed | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRI Group | Control Group | Total
Number analyzed (Participants) | 177 | 89 | 266
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.0 (10.4) | 67.8 (15.1) | 69.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 40 | 108
  Male | 109 | 49 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 52 | 26 | 78
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 87 | 45 | 132
  More than one race | 12 | 4 | 16
  Unknown or Not Reported | 26 | 14 | 40

OUTCOME MEASURES:

1. Primary Outcome: MRI-related Complication Free Rate
Description: Number of patients free of MRI-related complications
Time Frame: MRI scan to one month later
Population: Patients who underwent an MRI
Measure: Number; unit: participants
Arm/Group | MRI Group
Number analyzed (Participants) | 156
participants | 156
Statistical Analysis 1: Comparison: MRI Group; Null Hypothesis: MRI-related complication-free rate between the MRI scan and one-month post-MRI <90%; Test type: Superiority or Other; p < 0.0001, exact test of binomial proportions — A priori threshold for statistical significance was 0.025; Percentage = 100, 97.5% CI 1-sided [lower limit 97.7]

2. Primary Outcome: Proportion of Subjects Who Experience an Increase Less Than or Equal to 0.5V in Atrial Voltage Thresholds
Description: Subjects' atrial pacing capture threshold was measured at the 9-12 week visit (pre-MRI/waiting period) and the 4-month visit (i.e. one month post-MRI/waiting period). A success was when a subject experienced an increase less than or equal to 0.5V (volts) between the two visits.
Time Frame: Pre-MRI/waiting period (9-12 weeks post implant) to one month post-MRI/waiting period
Population: To be included in the analysis, subjects in the MRI group must undergo an MRI scan and those in the Control group must complete the 9-12 week visit, and all the subjects must have valid pacing capture threshold measurements at pre-MRI/waiting period and the 4-month visit.
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 142 | 80
participants | 142 | 80
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: % successes MRI group ≤ % successes Control group -10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; Farrington-Manning test — A priori threshold for statistical significance was 0.025. Because there were no failures in either group, a p-value could not be calculated; Risk Difference (RD) = 0

3. Primary Outcome: Proportion of Subjects Who Experience an Increase Less Than or Equal to 0.5V in Ventricular Voltage Thresholds
Description: Subjects' ventricular pacing capture threshold was measured at the 9-12 week visit (pre-MRI/waiting period) and the 4-month visit (i.e. one month post-MRI/waiting period). A success was when a subject experienced an increase less than or equal to 0.5V (volts) between the two visits.
Time Frame: Pre-MRI/waiting period (9-12 weeks post implant) to one month post-MRI/waiting period
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 153 | 82
participants | 152 | 82
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: % successes MRI group ≤ % successes Control group -10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; p < 0.0001, Farrington-Manning test — A priori threshold for statistical significance was 0.025; Risk Difference (RD) = -0.7, 95% CI 2-sided [-5.4 to 4.1]

4. Secondary Outcome: Proportion of Subjects Who Experience a Decrease Less Than or Equal to 50% in Atrial Sensing Amplitude
Description: Subjects' atrial sensed amplitude was measured at the 9-12 week visit (pre-MRI/waiting period) and the 4-month visit (i.e. one month post-MRI/waiting period). A success was defined as a 50% or less decrease in atrial sensed amplitude between the two visits.
Time Frame: Pre-MRI /waiting period (9-12 weeks post-implant) to 1-month post-MRI/waiting period
Population: Only subjects with measured sensed amplitude values at both pre-MRI/waiting period and the 4-month visit were used in the analysis.
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 144 | 81
participants | 141 | 78
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: % successes MRI group ≤ % successes Control group - 10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; p < 0.0001, Farrington-Manning test — A priori threshold for statistical significance was 0.05; Risk Difference (RD) = 1.6, 95% CI 1-sided [lower limit -3.2]

5. Secondary Outcome: Occurrence of Sustained Ventricular Arrhythmias and Asystole During MRI Scans.
Description: The endpoint was the occurrence of sustained ventricular arrhythmias and asystole during MRI scans and attributable to the MR scan. Sustained ventricular arrhythmias or asystole episodes that occurred during the MRI scan was considered attributable to the MR scan if so adjudicated by the Adverse Events Adjudication Committee
Time Frame: During MRI scans (9-12 weeks post-implant)
Measure: Number; unit: participants
Arm/Group | MRI Group
Number analyzed (Participants) | 159
participants | 0
Statistical Analysis 1: Comparison: MRI Group; Null hypothesis: the proportion of subjects with sustained ventricular arrhythmias and asystole during MRI scans >= 10%; Test type: Superiority or Other; p < 0.0001, exact test of binomial proportions; A priori threshold for statistical significance was 0.05; Percentage = 0, 95% CI 1-sided [upper limit 1.9]

6. Secondary Outcome: Proportion of Subjects Who Experience a Decrease Less Than or Equal to 50% in Ventricular Sensing Amplitude
Description: Subjects' ventricular sensed amplitude was measured at the 9-12 week visit (pre-MRI/waiting period) and the 4-month visit (i.e. one month post-MRI/waiting period). A success was defined as a 50% or less decrease in ventricular sensed amplitude between the two visits.
Time Frame: Pre-MRI/waiting period (9-12 weeks post implant) to one month post-MRI/waiting period
Measure: Number; unit: participants
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 139 | 79
participants | 134 | 76
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Null hypothesis: % successes MRI group ≤ % successes Control group - 10%; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was 10%; p = 0.0004, Farrington-Manning test; A priori threshold for statistical significance was 0.05; Risk Difference (RD) = 0.2, 95% CI 1-sided [lower limit -4.8]

ADVERSE EVENTS:
Time Frame: Implant to six-months post-implant
Arm/Group | MRI Group | Control Group
Serious Adverse Events (participants affected / at risk) | 28/177 | 6/89
Other Adverse Events (participants affected / at risk) | 0/177 | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Group (N=177) | Control Group (N=89)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 6 (6) | 0 (0)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Femoral Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Device Dislocation (General disorders) | 2 (2) | 2 (2)
Device Lead Issue (General disorders) | 1 (1) | 0 (0)
Device Pacing Issue (General disorders) | 1 (1) | 2 (2)
Implant Site Haematoma (General disorders) | 1 (1) | 0 (0)
Local Swelling (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood Sodium Decreased (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Medical Device Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No